CLINICAL TRIAL: NCT03795675
Title: Cochlear Implantation During Vestibular Schwannoma Removal or During Labyrinthectomy Surgery for Treatment of Meniere's Disease
Brief Title: CI Following VS Removal or Labyrinthectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Advanced Bionics (Industry)
Responsible Party: Principal Investigator, Oliver Adunka, Professor-Clinical Otolaryngology, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0273
Record Dates: First submitted 2018-12-07; First posted 2019-01-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Schwannoma; Meniere Disease
Keywords: Cochlear implants
MeSH Terms: conditions — Neuroma, Acoustic; Meniere Disease | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Meniere's Disease/Vestibular Schwannoma (Experimental): Individuals diagnosed with Meniere's disease and undergoing labyrinthectomy or diagnosed with vestibular schwannoma and undergoing surgical excision via translabyrinthine approach for treatment will receive cochlear implant at the time of surgery.
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — Cochlear implant device to be implanted at time of surgical intervention.

SUMMARY:
This study is a prospective, clinical study to determine if it is safe and effective to use a cochlear implant over time in individuals undergoing removal of a vestibular schwannoma (VS), benign tumor of the hearing and balance nerve or undergoing a labyrinthectomy for treatment of Meniere's disease. Individuals undergoing these surgeries will be deaf on the surgical side after the procedure. Currently, cochlear implants are approved for use and not considered investigational in individuals with hearing loss on both sides. However, use of a cochlear implant for these patient populations (single-sided hearing loss) will be considered a new use of an approved device. Participants undergoing surgery to remove a VS or having a labyrinthectomy will have a cochlear implant inserted after the surgical procedure for clinical care. Approximately 4 weeks after surgery, participants will be fitted with an external speech processor on the surgical side that will stimulate the internal cochlear implant. Participants will return at the following intervals after the initial processor fitting: 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months. At each interval, participants will complete questionnaires on how they are hearing with the implant and their quality of life with the implant and be tested on their ability to hear sounds and understand speech. Potential risks are those associated with all cochlear implant surgeries, and include device failure resulting in removal of device, irritation or redness in surgical area and/or area where processor is attached, increased ringing in the ear, facial nerve stimulation and a change in the way speech and other sounds sound through the implant. Potential benefits to individual participants in this study include improvement in detection and speech understanding of the surgical ear. Participants may also experience improved abilities to locate sound and understand speech in noise as the result of having hearing on both sides.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of a vestibular schwannoma confirmed by a physician with an MRI and/or CT scan; Or have a diagnosis of Meniere's disease by a physician
* Be scheduled to undergo surgery to remove the vestibular schwannoma through translabyrinthine approach; Or be scheduled to undergo a labyrinthectomy
* Be English-speaking due to objective speech perception tasks. Non-English speakers may show a reduced speech perception score due to language differences
* For patients undergoing tumor removal, tumor removal must allow preservation of the auditory division of the VIIIth cranial nerve

Exclusion Criteria:

* Subjects with bilateral Meniere's disease or bilateral vestibular schwannomas
* Inability to preserve the auditory division of the VIIIth cranial nerve during removal of vestibular schwannoma
* Ossification or fibrosis of the cochlear found on preoperative imaging (CT or MRI) that precludes cochlear implantation
* Active middle ear disease
* Greater than 70 years of age
* Vestibular schwannoma greater than 2 cm
* Patient refusal of receiving pneumococcal vaccine
* Any contra-indication(s) for undergoing surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-01-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Sound Detection Testing | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Sounds that vary in pitch (frequency) will be presented in a sound field to identify hearing thresholds in decibels (dB). Participant indicates when a sound is detected/perceived when listening with the cochlear implant. The softest sound at each specific frequency (125, 250, 500, 1000, 2000, 3000, 4000, 6000, 8000 Hertz (Hz)) will be recorded in dB hearing level.
Change in Speech Perception Testing | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Arizona (AZ) Bio sentences (speech perception test comprised of 660 unique sentences, presented in 33 independent lists of 20 sentences each) and the Maryland consonant-vowel nucleus-consonant (CNC) (10 phonetically balanced 50-word lists) word lists will be presented through a sound field speaker, and participant will be asked to repeat back the sentences and/or word that was heard. Background noise will be presented in conjunction with the sentences/words at various signals to noise levels (quiet [no noise], +0 dB and +5 dB signal to noise ratio). The percentage of sentences/words correctly repeated will be calculated for each test (AZ Bio, CNC) at each signal to noise level. Higher percentages indicate better word and sentence recognition ability.
Change in Sound Localization Testing | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Participant listens to bursts of sounds (100 trials of pink noise [random noise having equal energy per octave and having more low-frequency components than white noise; the power per hertz decreases as the frequency increases] presented randomly from seven speakers in a half-moon orientation and identifies which speaker presented the sounds. Two testing conditions will be evaluated (implant on, implant off). Total percentage of sounds correctly identified for each condition (0-100%) will be calculated, with a larger percentage indicating higher accuracy. Additionally, root mean square error (average of total degree of error when localizing) will be calculated for each trial.

SECONDARY OUTCOMES:
Change in Speech, Spatial and Qualities of Hearing Scale (SSQ) Scores | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Subjective questionnaire designed to study the relationship of disability and handicap across many listening domains using 49 questions in a clinician/patient interview format. The scale is sub-divided into three domains: 14 items on speech hearing, 17 items on spatial hearing (direction and distance judgments), and 18 items on "other" functions and qualities of hearing. The "other" qualities section contains items related to recognition and segregation of sounds, clarity, naturalness, and listening effort. Items are scored with ratings of 0 to 10, with 0 representing complete inability with regard to the item in question and 10 representing perfect ability. The average score (0-10) for each subscale/domain is reported individually.
Change in Nijmegen Cochlear Implant Questionnaire (NCIQ) Scores | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Questionnaire encompassing hearing and speech, psychological, and social domains and is used to evaluate quality of life. This questionnaire contains six subdomains of hearing that are rated categorically (1-5 (never-always) and "not applicable"). The subdomains are 1. Basic sound perception, 2. Advanced sound perception (in difficult daily listening situations or background noise), 3. Speech production, 4. Self-esteem, 5. Activity limitations, 6. Social interaction. The answer categories must first be transformed (1=0, 2=25, 3=50, 4=75 and 5=100). Afterwards, the final subdomain score is computed by adding together all the item scores and dividing by the number of completed items, resulting in a range of scores from 0 to 100. A higher score reflects a greater ability.
Change in Tinnitus Handicap Inventory (THI) Scores | Measurements assessed 2 weeks, 1 month, 3 months, 6 months, 9 months, and 12 months post-implantation.
  Subjective questionnaire that identifies, qualifies, and evaluates the difficulties that may be experienced due to tinnitus. It is a 25-item questionnaire grouped into three subscales: functional, emotional and catastrophic responses. The functional subscale items reflect the effect of tinnitus on mental, social, occupational and physical functioning. The emotional subscale items probe the individual's emotional reactions to tinnitus, and the catastrophic response items address whether tinnitus makes the respondent feel desperate, trapped, hopeless or out of control. A "yes" response is given 4 points, a "sometimes" response 2 points and a "no" response 0 points. The questionnaire yields scores for each subscale and a total score that ranges from 0 and 100, with high scores indicating a greater handicap. The total score of this questionnaire represents the overall severity of tinnitus: slight (0-16), mild (18-36), moderate (38-56), severe (58-76) or catastrophic (78-100).

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Adunka, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03795675/Prot_SAP_000.pdf